CLINICAL TRIAL: NCT06807658
Title: Cardiac Telerehabilitation Versus In-person After Acute Coronary Syndrome: Randomized Clinical Trial TELECOR Study
Brief Title: Cardiac Telerehabilitation Versus In-person After Acute Coronary Syndrome
Acronym: TELECOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PI-21-286; PI-21-286 (Other: Germans Trias i Pujol Ethics Committee)
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Acute Myocardial Infarction (AMI); Cardiac Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-rehabilitation (Experimental): Patients with a myocardial infarction candidates to a rehabilitation program, will be enrolled. The patient is guided via a face-to-face telematic call to perform the cardiac rehabilitation exercises and life style education.
  Interventions: Behavioral: Experimental: Cardiac tele-rehabilitation
- In person cardiac rehabilitation (Active Comparator): Patients with a myocardial infarction candidates to a rehabilitation program, will be enrolled. The patient attends an in-person cardiac rehabilitation exercises and life style education at the hospital.
  Interventions: Behavioral: Other: Control, in person cardiac rehabilitation

INTERVENTIONS:
Behavioral: Experimental: Cardiac tele-rehabilitation — Patients will connect to their health care provider via a tele-call
  Arms: Tele-rehabilitation
Behavioral: Other: Control, in person cardiac rehabilitation — Patients will attend an ambulatory cardiac rehabilitation unit
  Arms: In person cardiac rehabilitation

SUMMARY:
The purpose of this trial is to evaluate wether a cardiac Telerehabilitation programme is as effective as an in-person rehabilitation program after acute coronary syndrome in the control of cardiovascular risk factors

DETAILED DESCRIPTION:
The purpose of this trial is to evaluate wether a cardiac Telerehabilitation programme is as effective as an in-person rehabilitation program after acute coronary syndrome in the control of cardiovascular risk factors via the following variables: % patients with a positive result in the composite variable integrating different targets for secondary prevention in cardiovascular disease and lifestyle habits; Adherence to cardiac rehabilitation program; Adherence to pharmacological treatment; Quality of Life improvement ; Anxiety and depression; Satisfaction rate; Functional capacity; Cardiac cause hospitalization; Emergency visits; and Angioplasty revascularization procedure.

ELIGIBILITY:
Inclusion Criteria:

* Acute myocardial infarct prior to 2 months
* Killip I-II classification
* No previous myocardial infarction
* No angina pectoris
* No ischemia in complementary explorations
* Normal arterial pressure response during stress test.
* No relevant arrythmias
* Left ventricular ejection fraction >= 35%
* Functional capacity >5 METS
* Signing of the inform consent

Exclusion Criteria:

* Physical or intellectual disability that prevents patients from enrolling in a cardiac rehabilitation program
* Impossibility for digital media use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-02-02 (Actual)

PRIMARY OUTCOMES:
% patients with a positive result in the composite variable integrating different targets for secondary prevention in cardiovascular disease and lifestyle habits | • (%) [Time Frame: 0-2months +- 30 days-6 months +-7days]
  Variable for Cardiovascular Risk Factor Control: Composite Variable Integrating Different Targets for Secondary Prevention in Cardiovascular Disease and Lifestyle Habits
  1. Blood pressure <140/90 mmHg
  2. Maintaining normal weight or a 5% reduction in body weight if BMI > 25 kg/m2
  3. Abdominal circumference <88 cm in women and <102 cm in men
  4. LDL <50 mg/dl and a reduction of >50% in initial LDL levels
  5. Smoking cessation
  6. Adherence to a heart-healthy diet (PREDIMED Questionnaire* ≥7)
  7. Adherence to physical activity level: 6,000-10,000 steps/day or moderate-high IPAQ** result (International Physical Activity Questionnaire)

SECONDARY OUTCOMES:
Adherence to cardiac rehabilitation program | 2 months +-30 day
  % of patients adherent to cardiac rehabilitation program
Adherence to pharmacological treatment | 0-2months +- 30 days-6 months +-7days
  Adherence to pharmacological treatment by Morinsky Green Questionnaire, Dichotomous variable: yes means adherent to treatment wich is a better score and no means non adherent to treatment wich is a worse score.
Quality of Life improvement | 0-2months +- 30 days-6 months +-7days
  Quality of Life by EuroQol-5D questionnaire. EuroQoL-5D index (0-1) 0: Represent the worse state of Health, equivalent to death.
  1: Represents the best state of Health ( no problems in any dimension of the questionnaire).
Anxiety and depression | 0-2months +- 30 days-6 months +-7days
  Anxiety and depression by Hospital Anxiety and Depression Scale (HADS). HAD Questionnaire:
  0-42: Higher values are worse than lower values.
Satisfaction rate | 2months +- 30 days
  Satisfaction rate with the program, Scale 0-100 (%); 0-100%: Higher values are better than lower values
Functional capacity | 0-2months +- 30 days
  Functional capacity by cardiac stress test (METS)
Cardiac cause hospitalization | 6 months +-7days
  Cardiac cause hospitalization
Emergency visits | 6 months +-7days
  Emergency visits
Angioplasty revascularization procedure | 0-2months +- 30 days
  Angioplasty revascularization procedure. Further coronary angiography during follow up Yes: is worse No: is better

OTHER OUTCOMES:
Cost analysis | 6 months +-7days
  Analyze in terms of economic cost (euros) whether there are differences between both programs ( total cost of Telerehabilitation program and total cost of in person program) Total cost includes: direct costs, indirect costs, and intangible costs.

CONTACTS AND LOCATIONS:
Locations (1):
- Germans Trias i Pujol University Hospital, Badalona, Spain

IPD SHARING:
Plan to Share IPD: Undecided